CLINICAL TRIAL: NCT03697317
Title: Televideo Exercise and Nutrition Program for Kidney Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Cheryl Gibson, Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00140695
Record Dates: First submitted 2018-09-21; First posted 2018-10-05 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Kidney Transplant Recipient; Diet Modification; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Televideo Lifestyle Coaching (Experimental)
  Interventions: Behavioral: Televideo Lifestyle Coaching
- Enhanced Usual Care (Active Comparator)
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Televideo Lifestyle Coaching — Six month total intervention: Three months of weekly 1-hour televideo healthy lifestyle coaching sessions involving 30 minutes of structured physical activity and 30 minutes of nutrition education and daily healthy lifestyle habit tracking. This is followed by 3 months of healthy lifestyle habit tracking only.
  Arms: Televideo Lifestyle Coaching
Behavioral: Enhanced Usual Care — Six months of healthy lifestyle habit tracking with access to written diet and physical activity materials.
  Arms: Enhanced Usual Care

SUMMARY:
The improvement in morbidity and mortality observed with kidney transplantation is often curtailed by post-transplant weight gain, which is common among kidney transplant recipients (KTR). Post-transplant weight gain is associated with serious health issues such as cardiovascular disease, new onset diabetes after transplantation, and graft failure. Although these adverse effects of post-transplant weight gain are well recognized, interventions that target the modifiable risk factors of diet and physical activity to address post-transplantation weight gain are lacking. The purpose of this study is to test the feasibility of an in-home, televideo health coaching to increase the healthy behaviors of KTRs who are 6 months post-transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Between 6 and 12 months post kidney transplantation
* Kidney allograft only
* Functioning allograft (not on dialysis)
* BMI ≥ 22 kg/m2
* Available to participate in assessments over 6 months
* Ability to speak and understand English
* Able to report data weekly by at least one of three alternative methods: telephone, email, or fax
* Access to wireless internet

Exclusion Criteria:

* Multi-organ transplant recipient
* Uncontrolled diabetes (Hemoglobin A1c≥8%)
* Currently pregnant or planning on becoming pregnant during the study
* Participation in a formal weight management, nutrition, or physical activity program
* Diagnosis of a major psychiatric illness
* Major dietary restrictions
* Inability to perform moderate to vigorous physical activity
* Unwillingness to be randomized
* Receiving supplemental nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Recruitment of participants | 1 month
  Achievement of 10 participants in 1 months
Attendance to group sessions | 3 months
  Maintain 80% attendance or better to program sessions
Participant retention in study assessments | 6 months
  85% or greater participant retention in study assessments

SECONDARY OUTCOMES:
Change in diet quality assessed by Healthy Eating Index Scores | Change from baseline to month 6
  Changes in dietary quality will be determined by calculating Healthy Eating Index- 2010 scores from 3 day food records. A total HEI-2010 score will be calculated, which is comprised of a summative score across 12 subscales, with higher scores indicative of a better diet quality (maximum score 100).
Change in weight | Change from baseline to month 6
  Weight in kilograms will be measured with a digital scale

OTHER OUTCOMES:
Quality of Life-Kidney Transplant Questionnaire (KTQ) | Baseline, 3 months, 6 months
  Quality of life will be assessed using the Kidney Transplant Questionnaire, a 25-question disease-specific questionnaire with 5 dimensions measured- physical symptoms, fatigue, uncertainty/fear, appearance, and emotions. A higher score indicates a greater quality of life. A change in score greater than 0.5 in each domain is clinically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl A Gibson, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Gibson CA, Gupta A, Greene JL, Lee J, Mount RR, Sullivan DK. Feasibility and acceptability of a televideo physical activity and nutrition program for recent kidney transplant recipients. Pilot Feasibility Stud. 2020 Sep 10;6:126. doi: 10.1186/s40814-020-00672-4. eCollection 2020. PMID 32944274